CLINICAL TRIAL: NCT03280459
Title: Prospective Cohort-study for Evaluation of Clinical Outcome of Robot-assisted Cystectomy With Intracorporeal Reconstruction of Urinary Diversion
Brief Title: Evaluation of Robot-assisted Intracorporeal Urinary Reconstruction
Acronym: iRARC-KSW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Christoph Schregel, Assistenzarzt Urologie / resident Departement of Urology, Kantonsspital Winterthur KSW
Other Study IDs: 2017-01260
Record Dates: First submitted 2017-08-29; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Urothelial Carcinoma; Cystectomy; Urinary Diversion; Complication of Surgical Procedure; Complication, Postoperative; Neobladder; Ileal Conduit; Robotic Surgical Procedures
MeSH Terms: conditions — Carcinoma, Transitional Cell; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ileal Conduit: Patient with ileal conduit as reconstruction of urinary diversion after robot-assisted cystectomy
  Interventions: Procedure: robot-assisted cystectomy
- Neobladder: Patient with neobladder, (orthotopic, continent ileal pouch) as reconstruction of urinary diversion after robot-assisted cystectomy
  Interventions: Procedure: robot-assisted cystectomy

INTERVENTIONS:
Procedure: robot-assisted cystectomy — Removal of urinary bladder in oncologic or functional setting using a assistance of a operation robotic for laparoscopy

SUMMARY:
Continous evaluation of clinical and oncologic outcome of robot-assisted cystectomy with intracorporeal reconstruction of urinary diversion. Patient Data is entered in an anonymized registry for analyzation.

DETAILED DESCRIPTION:
The registry includes patients after robot-assisted cystectomy, mainly as therapy for muscle invasive urothelial carcinoma. The urinary diversion will be completed intracorporeal either as ileal conduit or ileal neobladder. Outcome parameters include perioperative complications, oncologic data and oncologic follow-up data (tumor classification, recurrence, survival) as well as data on functional follow up (continence, quality of life).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years
* informed consent for operation and data use
* Oncologic patients that qualify for radical cystectomy according to institutional tumor-board decision or patients with functional indications after failure of all other therapy modalities and receive a cystectomy

Exclusion Criteria:

* age <18 years
* declined informed consent / data use
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Onkologic patients that qualify for radical cystectomy according to institutional tumor-board decision or patients with functional indications after failure of all other therapy modalities and receive a cystectomy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 1 year
  deviations from normal postoperative course ["Clavien-Dindo" Grade]

SECONDARY OUTCOMES:
Treatment of tumor recurrence | through study completion, an average of 5 years
  Treatment of tumor recurrence (radiotherapy, chemotherapy, operation)
Quality of Life urology specific | 1 year
  EORTC-BLM 30 (European Organisation for Research and Treatment of Cancer Questionaire for muscle invasive bladder cancer) questionaire for evaluation of quality of life for patients with muscle invasive bladder cancer
Quality of Life overall | 1 year
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionaire) questionaire for evaluation of quality of life for oncologic patients
Operation Time | expected 4-8 hours
  duration of operation [min]
Postoperative Death by any cause | through study completion, an average of 5 years
  Death by any cause [n/months]
Pouch capacity | 1 year
  interventional measurement of pouch capacity with pressure recording catheter [ml]
Type of tumor-recurrence | through study completion, an average of 5 years
  Location of tumor recurrence (local, metastasis)
Blood loss | expected 4-8 hours
  blood loss during operation [ml]
Time to recurrence | through study completion, an average of 5 years
  time until recurrence of tumor [months]
Tumor specific death | through study completion, an average of 5 years
  Time to tumor specific death [months]
Preoperative Tumor staging | 90 days
  Preoperative Tumor staging according UICC TNM System (Union internationale contre le cancer Tumor Nodus Metastasis System)
Postoperative Tumor staging | 90 days
  Postoperative Tumor staging according UICC TNM System (Union internationale contre le cancer Tumor Nodus Metastasis System)
Pouch-pressure | 1 year
  interventional measurement of pouch-pressure [cmH2O]with pressure recording catheter
Postvoid residual urine | 1 year
  Residual urin after voiding [ml]
Functional length of urethral sphincter | 1 year
  interventional measurement of Functional length of urethral sphincter [mm] with pressure recording catheter
Functional pressure of urethral sphincter | 1 year
  interventional measurement of functional pressure of urethral sphincter [cmH2O] with pressure recording catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
depersonalized Data may be shared with other academic centers if data security and ethical considerations equal to swiss standards are followed